CLINICAL TRIAL: NCT02160652
Title: Ureteral Reimplantation for the Treatment of Extrinsic Malignant Ureteral Obstruction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0185-14-RMC
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Ureteral Obstruction
Keywords: Ureteral Obstruction; HYDRONEPHROSIS; nephrostomy tube
MeSH Terms: conditions — Ureteral Obstruction; Hydronephrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: Patients with malignant ureteral obstruction, treated with laparoscopic ureteral re-implantation, who have a life expectancy of over 6 months and are willing and able to participate in the study.
  Interventions: Procedure: Laparoscopic ureteral re-implantation.

INTERVENTIONS:
Procedure: Laparoscopic ureteral re-implantation. — Laparoscopic ureteral re-implantation for the treatment of malignant ureteral obstruction.

SUMMARY:
A single center single arm prospective study, assessing the outcome of ureteral re-implantation for malignant ureteral obstruction.

DETAILED DESCRIPTION:
The Research Question: Is laparoscopic ureteral re-implantation, for the treatment of malignant ureteral obstruction, associated with high patency rates, low complication rates, and a significant improvement in quality of life?

Study design: A single center single arm prospective study, assessing the outcome of ureteral re-implantation for malignant ureteral obstruction.

Study population: Patients with malignant ureteral obstruction, treated with laparoscopic ureteral re-implantation, who have a life expectancy of over 6 months and are willing and able to participate in the study.

Intervention: Laparoscopic ureteral re-implantation.

Study Time line: This will be a 1 year study. At initiation a baseline physical exam, blood test, and ultrasonography will be performed. Baseline quality of life questionnaires will be filled. After the operation, Follow-up visits will occur at 1, 3, 6 and 12 months after surgery. At each follow up visit a medical history and physical examination, blood tests and quality of life questionnaires will be performed. At 3, 6 and 12 months renal ultrasonography will be performed.

Primary Endpoint: Ureteral patency at 6 months following treatment - assessed by stable or improved hydronephrosis and estimated glomerular filtration rate (eGFR) according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

Study impact: Current treatments for malignant ureteral obstruction with nephrostomy tubes negatively impact the patient's quality of life. The findings of the current study may support the use of laparoscopic ureteral re-implantation for the treatment of malignant ureteral obstruction, if patency is preserved, and quality of life is improved, following the procedure.

ELIGIBILITY:
Inclusion criteria:

1. Adult patient, older than 18 years of age.
2. Patient with malignant ureteral obstruction diagnosed by creatinine elevation with evidence of ureteral obstruction on imaging.
3. Patient is scheduled for ureteral reimplantation due to extrinsic malignant ureteral obstruction.
4. American Society of Anesthesiologist score ≤3, enabling the patient to undergo surgery.
5. Life expectancy of over 6 months ( see exclusion criteria for definition)
6. WHO performance status 0-2
7. The patient is willing and able to read, understand and sign the study specific informed consent form

Exclusion criteria:

1. Patients who underwent urinary diversion other than percutaneous nephrostomy or retrograde ureteral stenting prior to the planned treatment.
2. Patients unable to sign an informed consent for or unwilling to undergo so.
3. Life expectancy of less than 6 months, as defined according to the criteria by Ishioka et al. and predicted in the presence of:

   * Low serum albumin before percutaneous nephrostomy/ retrograde ureteral stenting (3 gm/dl or less).
   * Low grade hydronephrosis prior to percutaneous nephrostomy/ retrograde ureteral stenting placement (grade 1 or 2) as graded by the grading system of the Society for Fetal Urology
   * Malignant ascites or malignant pleural effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant ureteral obstruction, treated with laparoscopic ureteral re-implantation, who have a life expectancy of over 6 months and are willing and able to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Ureteral patency - 6 months | 6 months following the operation
  Ureteral patency at 6 months following the operation- assessed by stable or improved hydronephrosis and estimated GFR according to the CKD-EPI equation.

SECONDARY OUTCOMES:
Ureteral patency - 12 months | 12 months following the operation
  Ureteral patency at 12 months following the operation.
Post-operative complications | 1, 3, 6, and 12-months following the operation
  Post-operative complications 1, 3, 6, and12-months following the operation
Quality of life | 1,3,6, and 12 months following the operation
  Changes in quality of life at 1,3, 6 and 12 months following the operation. Quality of life will be evaluated using two questionnaires:
  * Functional Assessment of Cancer Therapy scale - General (FACT-G).
  * Intervention specific questionnaire based on Joshi et al. ()
Re-intervention | 12 months following the operation
  Re-interventions following the operation.

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD, PhD, Principal Investigator — Rabin Medical Center

IPD SHARING:
Plan to Share IPD: Undecided